CLINICAL TRIAL: NCT03316976
Title: A Phase 1, Single-Center, Open-Label, 2-Arm Parallel Group, Single-Dose Study to Evaluate the Pharmacokinetics of Dexlansoprazole 30 mg and 60 mg Delayed-Release Capsules in Healthy Chinese Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics of Dexlansoprazole 30 Milligram (mg) and 60 mg Delayed-release Capsules in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAK-390MR_106; U1111-1192-7711 (Registry Identifier: WHO); CTR20160792 (Registry Identifier: SFDA)
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Results first posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-02

CONDITIONS: Healthy Volunteers
Keywords: Drug therapy
MeSH Terms: interventions — Dexlansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Dexlansoprazole 30 mg (Experimental): Dexlansoprazole 30 mg, delayed-release, capsule, orally, administered as single dose on Day 1.
  Interventions: Drug: Dexlansoprazole
- Group 2: Dexlansoprazole 60 mg (Experimental): Dexlansoprazole 60 mg, delayed-release, capsule, orally, administered as single dose on Day 1.
  Interventions: Drug: Dexlansoprazole

INTERVENTIONS:
Drug: Dexlansoprazole — Dexlansoprazole delayed-release capsule.
  Other Names: TAK-390 Modified Release (TAK-390MR) dexlansoprazole

SUMMARY:
The purpose of this study is to assess the pharmacokinetics after a single dose of dexlansoprazole 30 and 60 mg delayed-release capsules in healthy Chinese participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called Dexlansoprazole. This study will assess the pharmacokinetics, safety and tolerability of a single oral dose of Dexlansoprazole 30 mg and 60 mg delayed-release capsules in healthy participants.

The study will enroll approximately 40 participants, 20 participants in each parallel arm. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups:

* Group 1: A single oral dose of Dexlansoprazole 30 mg delayed-release capsule
* Group 2: A single oral dose of Dexlansoprazole 60 mg delayed-release capsule

All participants will be asked to take single dose of study drug on Day 1.

This single center trial will be conducted in China. The overall time to participate in this study is approximately 40 days. Participants will be contacted by telephone or will make a final visit to the clinic 5 to 10 days after receiving their last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy adult man or woman of Chinese descent.
2. Is aged 18 to 45 years, inclusive, at the time of informed consent and study medication dose.
3. Weighs at least 50 kilogram (kg) and has a body mass index (BMI) from 19.0 to 26.0 kilogram per square meter (kg/m^2), inclusive at Screening Visit.

Exclusion Criteria:

1. Has a known hypersensitivity to any component of the formulation of dexlansoprazole or other drug with the same mechanism of action (including lansoprazole, omeprazole, esomeprazole, rabeprazole, ilaprazole, or pantoprazole), or related compounds.
2. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to the Screening visit or is unwilling to agree to abstain from alcohol for 48 hours prior to Check-in (Day -1) throughout the confinement and for 48 hours prior to each clinic visit and drugs throughout the study.
3. Has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 28 days prior to Check-in (Day -1) or is unwilling to abstain from these products for the duration of the study.
4. Has poor peripheral venous access.
5. Has donated blood products (such as plasma), whole blood or had a significant blood loss (450 millimeter [mL]) within 56 days of Day 1.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2018-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Phase I Clinical Trial Department, Beijing, Beijing Municipality, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in China from 22 November 2017 to 08 February 2018.
Pre-assignment Details: Healthy Chinese participants were enrolled in this two arm study to receive single oral dose of dexlansoprazole 30 and 60 milligram (mg) delayed-release capsules.
Period: Overall Study
Arm/Group | Group 1: Dexlansoprazole 30 mg | Group 2: Dexlansoprazole 60 mg
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who were enrolled in the study and received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Dexlansoprazole 30 mg | Group 2: Dexlansoprazole 60 mg | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The safety analysis set included all participants who were enrolled in the study and received at least 1 dose of study drug.
  years | 29.4 (6.73) | 29.4 (5.66) | 29.4 (6.14)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The safety analysis set included all participants who were enrolled in the study and received at least 1 dose of study drug.
  Participants
    Female | 12 | 7 | 19
    Male | 8 | 13 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — Population: The safety analysis set included all participants who were enrolled in the study and received at least 1 dose of study drug.
  Participants
    China | 20 | 20 | 40
Height [Mean (Standard Deviation); unit: centimeter] — Population: The safety analysis set included all participants who were enrolled in the study and received at least 1 dose of study drug.
  centimeter | 165.88 (7.688) | 167.38 (7.720) | 166.63 (7.642)
Weight [Mean (Standard Deviation); unit: kilogram] — Population: The safety analysis set included all participants who were enrolled in the study and received at least 1 dose of study drug.
  kilogram | 61.22 (8.469) | 62.43 (8.542) | 61.82 (8.418)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — Population: The safety analysis set included all participants who were enrolled in the study and received at least 1 dose of study drug.
  kilogram per square meter (kg/m^2) | 22.17 (1.808) | 22.22 (1.911) | 22.20 (1.836)
Smoking Classification [Count of Participants; unit: Participants] — Population: The safety analysis set included all participants who were enrolled in the study and received at least 1 dose of study drug.
  Participants
    Never smoked | 15 | 17 | 32
    Ex-Smoker | 5 | 3 | 8
Caffeine Consumption Status 72 hours Prior to Check-in (Day -1) [Count of Participants; unit: Participants] — Population: The safety analysis set included all participants who were enrolled in the study and received at least 1 dose of study drug.
  Participants
    Had caffeine consumption | 0 | 0 | 0
    Had no caffeine consumption | 20 | 20 | 40
Alcohol Consumption Status 7 Days Prior to Check-in (Day -1) [Count of Participants; unit: Participants] — Population: The safety analysis set included all participants who were enrolled in the study and received at least 1 dose of study drug.
  Participants
    Had alcohol consumption | 0 | 0 | 0
    Had no alcohol consumption | 20 | 20 | 40
Drug Abuse/Addiction [Count of Participants; unit: Participants] — Population: The safety analysis set included all participants who were enrolled in the study and received at least 1 dose of study drug.
  Participants
    Had a history of drug abuse/addiction | 0 | 0 | 0
    Had no history of drug abuse/addiction | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Dexlansoprazole
Time Frame: Day 1 pre-dose and at multiple timepoints (up to 24 hours) post-dose
Population: The pharmacokinetics (PK) set included all participants who received at least 1 dose of study drug and had at least 1 measureable plasma concentration of dexlansoprazole.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Group 1: Dexlansoprazole 30 mg | Group 2: Dexlansoprazole 60 mg
Number analyzed (Participants) | 20 | 20
nanogram per milliliter (ng/mL) | 732 (43.73) | 1756 (45.83)

2. Primary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Dexlansoprazole
Time Frame: Day 1 pre-dose and at multiple timepoints (up to 24 hours) post-dose
Population: The PK set included all participants who received at least 1 dose of study drug and had at least 1 measureable plasma concentration of dexlansoprazole.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Group 1: Dexlansoprazole 30 mg | Group 2: Dexlansoprazole 60 mg
Number analyzed (Participants) | 20 | 20
hour*nanogram per milliliter (h*ng/mL) | 3660 (61.38) | 10198 (61.09)

3. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Dexlansoprazole
Time Frame: Day 1 pre-dose and at multiple timepoints (up to 24 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Group 1: Dexlansoprazole 30 mg | Group 2: Dexlansoprazole 60 mg
Number analyzed (Participants) | 20 | 20
h*ng/mL | 3701 (62.83) | 10340 (64.20)

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days after last dose (Day 31)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Group 1: Dexlansoprazole 30 mg | Group 2: Dexlansoprazole 60 mg
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 3/20 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Dexlansoprazole 30 mg (N=20) | Group 2: Dexlansoprazole 60 mg (N=20)
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
White blood cells urine (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/76/NCT03316976/SAP_000.pdf
  • Study Protocol (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/76/NCT03316976/Prot_001.pdf